CLINICAL TRIAL: NCT02317146
Title: A Novel Protocol for Postpartum Magnesium Sulfate in Severe Preeclampsia When the Woman Received Less That 8 Hours Before Delivery. Six Versus Twenty-four Hours Postpartum
Brief Title: Magnesium Sulfate in Pregnancy and Postpartum
Acronym: MAG-PP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Complejo Hospitalario Dr. Arnulfo Arias Madrid (Other)
Responsible Party: Principal Investigator, Paulino Vigil-De Gracia, Co-Investigator, Complejo Hospitalario Dr. Arnulfo Arias Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: complejoh4
Record Dates: First submitted 2014-12-11; First posted 2014-12-15 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Severe Pre-eclampsia With Postnatal Complication
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Six Hours Postpartum (Experimental): The woman received magnesium sulfate for 6 hours after delivery as prophylaxis to eclampsia.
  Interventions: Drug: Magnesium Sulfate
- Twenty-four hours Postpartum (Active Comparator): The woman received magnesium sulfate for 24 hours after delivery as prophylaxis to eclampsia.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Magnesium sulfate is the drug used as prophylaxis to eclampsia in women with severe preeclampsia
  Other Names: anticonvulsivant

SUMMARY:
There are huge doubts as to how long to keep postpartum magnesium sulfate. Studies demonstrating the usefulness for 24, 12 or 6 hours are of little evidence and do not take into account the use of magnesium sulphate before delivery. Termination of pregnancy is the best option to prevent eclampsia and magnesium sulphate has proven effective, but do not know the minimum effective dose.The investigators believe that if the patient has received less than 8 continuous hours of magnesium sulphate before delivery, maintain magnesium sulfate for 6 hours is as effective as keeping it for 24 hours.

DETAILED DESCRIPTION:
The definitive treatment known for pre-eclampsia is the interruption of pregnancy. While the definitive treatment is the pregnancy interruption, management includes other measures that have proven effective, including the administration of antihypertensive drugs for severe hypertension and that the use of anticonvulsant such as the magnesium sulfate.

There are multiple studies that prove the effectiveness of magnesium sulfate to prevent eclampsia in patients with severe / serious disorder. Unfortunately these studies used the drug before birth and continue after birth. Therefore the investigators can not conclude whether the administration just before pregnancy is sufficient to prevent seizure. That is, if the cure or definitive treatment of pre-eclampsia is the interruption, did not seem necessary to justify the administration of anticonvulsant drugs after birth. Obvious post delivery management sulfate arises from the large number of postpartum eclampsia reported in many studies. It is unknown if the administration of magnesium sulfate for a minimum period not yet determined before birth and delivery requires even keep the drug after discontinuation.

For all these reasons the investigators propose the following: A randomized trial where all those patients who received magnesium sulfate for less that 8 hours before birth will be randomized to two groups of study: 1- Continue magnesium sulfate for 24 hours and 2-Continue magnesium sulfate for 6 hours postpartum.

ELIGIBILITY:
Inclusion Criteria:

Severe hypertensive disorder receiving magnesium sulfate prophylaxis for less than 8 hours at birth.

Exclusion Criteria:

* Complications such as: HELLP syndrome, renal failure, eclampsia, retinal detachment, cerebral edema, pulmonary edema, hypertensive encephalopathy.

Ages: 14 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 280 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Seizure (Eclampsia) | 72 hours postpartum
  Seizure during the first 72 hours post delivery

SECONDARY OUTCOMES:
Diuresis postpartum | 72 hours postpartum
  volume of urine post delivey
Persistent symptomatology | 24 hours postpartum
  headache, epigastric pain, visual and auditory symptoms symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Lewis, MD, Principal Investigator — Caja de seguro Social
Locations (3):
- Panama (3):
  - Hospital Jose Domingo de Obaldia, Chiriquí, Chiriquí Province
  - Hospital Manuel Amador Guerrero, Colón, Provincia de Colón
  - Complejo Hospitalario Caja de Seguro Social, Panama City, Provincia de Panamá

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altman D, Carroli G, Duley L, Farrell B, Moodley J, Neilson J, Smith D; Magpie Trial Collaboration Group. Do women with pre-eclampsia, and their babies, benefit from magnesium sulphate? The Magpie Trial: a randomised placebo-controlled trial. Lancet. 2002 Jun 1;359(9321):1877-90. doi: 10.1016/s0140-6736(02)08778-0. PMID 12057549
- [Background] Ascarelli MH, Johnson V, May WL, Martin RW, Martin JN Jr. Individually determined postpartum magnesium sulfate therapy with clinical parameters to safely and cost-effectively shorten treatment for pre-eclampsia. Am J Obstet Gynecol. 1998 Oct;179(4):952-6. doi: 10.1016/s0002-9378(98)70195-4. PMID 9790377
- [Background] Belfort MA, Anthony J, Saade GR, Allen JC Jr; Nimodipine Study Group. A comparison of magnesium sulfate and nimodipine for the prevention of eclampsia. N Engl J Med. 2003 Jan 23;348(4):304-11. doi: 10.1056/NEJMoa021180. PMID 12540643
- [Derived] Diaz V, Long Q, Oladapo OT. Alternative magnesium sulphate regimens for women with pre-eclampsia and eclampsia. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD007388. doi: 10.1002/14651858.CD007388.pub3. PMID 37815037
- [Derived] Vigil-De Gracia P, Ramirez R, Duran Y, Quintero A. Magnesium sulfate for 6 vs 24 hours post delivery in patients who received magnesium sulfate for less than 8 hours before birth: a randomized clinical trial. BMC Pregnancy Childbirth. 2017 Jul 24;17(1):241. doi: 10.1186/s12884-017-1424-3. PMID 28738788